CLINICAL TRIAL: NCT03567382
Title: Arresting Vertical Transmission of Hepatitis B Virus in the Democratic Republic of the Congo: The AVERT-HBV Study
Brief Title: Arresting Vertical Transmission of Hepatitis B Virus
Acronym: AVERT-HBV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Kinshasa School of Public Health (Other); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-2090; IGHID 11720 (Other: UNC Institute for Global Health and Infectious Diseases)
Record Dates: First submitted 2017-09-13; First posted 2018-06-25 (Actual); Results first posted 2021-02-05 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis B; Vertical Transmission of Infectious Disease
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir; Engerix-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- High-risk HBV dyads (Experimental): Mothers with high-risk HBV (defined as viral load >10^6 and/or HBeAg positivity) will be treated with tenofovir disoproxil fumarate (TDF) to further reduce the risk of vertical transmission of HBV. All HBV-exposed infants (regardless of mother's status of high- or low-risk HBV) will receive monovalent HBV vaccine within 24 hours of life.
  Interventions: Drug: Tenofovir Disoproxil Fumarate; Biological: Monovalent HBV vaccine
- Low-risk HBV dyads (Experimental): Mothers with low risk HBV (defined as a viral load <10^6 and negative HBeAg) will not receive tenofovir disoproxil fumarate therapy during or after pregnancy. Their infants will still receive monovalent HBV vaccine within 24 hours of life.
  Interventions: Biological: Monovalent HBV vaccine

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — 300 mg tablet of TDF once daily from 28-32 weeks gestation through 12 weeks postpartum.
  Other Names: Viread
  Arms: High-risk HBV dyads
Biological: Monovalent HBV vaccine — Infants born to HBsAg-positive women will be given a single dose of monovalent HBV vaccine within 24 hours of life.
  Other Names: Engerix-B

SUMMARY:
The purpose of this pilot study is to demonstrate the feasibility of adding HBV screening and treatment of pregnant women to the existing HIV PMTCT platform in order to prevent mother-to-child transmission of hepatitis B virus.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) is a leading cause of chronic liver disease globally, with devastating complications such as cirrhosis, hepatocellular carcinoma and death. Vertical transmission (VT) of HBV is a worldwide public health concern because infected children are at high risk of developing chronic liver disease. It is a particular problem in the Democratic Republic of the Congo (DRC); preliminary data suggest that approximately 3% of children have HBV infection due to VT. However, VT is preventable. Pregnant women with risk factors can be identified and treatments given which can virtually eliminate transmission. Unfortunately, despite the high burden of HBV, neither HBV testing of pregnant women nor interventions to prevent HBV VT are routinely performed in the DRC and elsewhere in sub-Saharan Africa. This pilot feasibility study will address this healthcare gap by identifying women with HBV early in their pregnancies and intervening to prevent VT by (1) treating mothers with high-risk HBV (defined as HBeAg positivity and/or HBV viremia >10^6) with tenofovir and (2) providing HBV vaccine to HBV-exposed infants within 24 hours of birth. This pilot study will piggyback onto an existing study that is evaluating the DRC's HIV Prevention of Maternal-to-Child Transmission Option B+ (PMTCT+) strategy. Combining programs to prevent VT of HBV and HIV enables using the same personnel and infrastructure to implement both interventions. Furthermore, tenofovir, used to treat HBV infections, is already used in the DRC to treat HIV. Researchers hypothesize that utilizing the existing PMTCT+ infrastructure in the DRC will provide a cost-effective platform to prevent HBV VT. If effective, this model of treatment will inform future public health efforts and wider policy recommendations that can be applied in the DRC and throughout the Sub-Saharan African region to reduce the burden of HBV.

ELIGIBILITY:
Inclusion criteria:

* Pregnant women receiving care at Binza and Kingasani maternity centers presenting prior to 24 weeks gestation
* Infants born to HBV-positive women

Exclusion criteria:

* Participants who are severely sick and who require prolonged hospitalization.
* Any women who do not intend to stay in Kinshasa for prenatal care through delivery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Meshnick, MD, Study Director — University of North Carolina, Chapel Hill; Peyton Thompson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Kinshasa School of Public Health, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thompson P, Morgan CE, Ngimbi P, Mwandagalirwa K, Ravelomanana NLR, Tabala M, Fathy M, Kawende B, Muwonga J, Misingi P, Mbendi C, Luhata C, Jhaveri R, Cloherty G, Kaba D, Yotebieng M, Parr JB. Arresting vertical transmission of hepatitis B virus (AVERT-HBV) in pregnant women and their neonates in the Democratic Republic of the Congo: a feasibility study. Lancet Glob Health. 2021 Nov;9(11):e1600-e1609. doi: 10.1016/S2214-109X(21)00304-1. Epub 2021 Aug 17. PMID 34416175

RESULTS

PARTICIPANT FLOW:
Groups:
- High-risk Mothers: Mothers with high-risk HBV (defined as viral load >10^6 and/or HBeAg positivity) will be treated with tenofovir disoproxil fumarate (TDF) to further reduce the risk of vertical transmission of HBV. All HBV-exposed infants (regardless of mother's status of high- or low-risk HBV) will receive monovalent HBV vaccine within 24 hours of life.
  Tenofovir Disoproxil Fumarate: 300 mg tablet of TDF once daily from 28-32 weeks gestation through 12 weeks postpartum.
  Monovalent HBV vaccine: Infants born to HBsAg-positive mothers will be given a single dose of monovalent HBV vaccine within 24 hours of life.
- Low-risk Mothers: Mothers with low risk HBV (defined as a viral load <10^6 and negative HBeAg) will not receive tenofovir disoproxil fumarate therapy during or after pregnancy. Their infants will still receive monovalent HBV vaccine within 24 hours of life.
  Monovalent HBV vaccine: Infants born to HBsAg-positive mothers will be given a single dose of monovalent HBV vaccine within 24 hours of life.
- Infants Born to High-risk Mothers: Infants born to mothers with high-risk HBV
- Infants Born to Low-risk Mothers: Infants born to mothers with low-risk HBV
Period: Overall Study
Arm/Group | High-risk Mothers | Low-risk Mothers | Infants Born to High-risk Mothers | Infants Born to Low-risk Mothers
Started | 10 | 81 | 9 | 79
Received Tenofovir | 9 | 0 | 0 | 0
Completed | 7 | 46 | 7 | 46
Not Completed | 3 | 35 | 2 | 33
Not completed — Lost to Follow-up | 1 | 21 | 1 | 21
Not completed — Withdrawal by Subject | 2 | 14 | 1 | 12

BASELINE CHARACTERISTICS:
Population: Baseline data were not collected for the Infant Arm/Groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | High-risk Mothers | Low-risk Mothers | Total
Number analyzed (Participants) | 10 | 81 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.4 (5.4) | 30.59 (5.47) | 29.91 (5.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 81 | 91
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Congo, The Democratic Republic of the | 10 | 81 | 91
Gestational age at enrollment, Continuous [Mean (Standard Deviation); unit: weeks] | 20.8 (3.55) | 17.54 (4.65) | 17.91 (4.64)
Total pregnancies, Continuous [Mean (Standard Deviation); unit: pregnancies] | 2.7 (2.06) | 3.52 (2.01) | 3.43 (2.02)
Number of living children, Continuous [Mean (Standard Deviation); unit: living children] | 0.89 (1.54) | 2.25 (1.80) | 2.10 (1.82)
Marital status, Categorical [Count of Participants; unit: Participants]
  Married | 7 | 66 | 73
  Divorced | 0 | 1 | 1
  Separated | 0 | 1 | 1
  Never Married | 2 | 13 | 15
  Missing | 1 | 0 | 1
Highest Education, Categorical [Count of Participants; unit: Participants]
  Primary | 1 | 1 | 2
  Secondary | 6 | 59 | 65
  Higher education | 3 | 17 | 20
  Missing | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Lab Testing Acceptability Survey Scores >80%
Description: The acceptability of laboratory testing approach to participants will be defined as >80% acceptability on a two questions each measured using a 5-point Likert scale (range 1-5, highest score of 5 representing the highest acceptability). For example, the options for participant responses will include: "Very unacceptable" (1), "Somewhat unacceptable" (2), "No opinion" (3), "Somewhat acceptable" (4), "Very acceptable" (5) and "Did not allow study personnel to take my blood". Scores equal to or greater than 4 considered 80%.
Time Frame: Upon completion of the exit survey, or up to 12 months
Population: There were a total of 53 mothers (7 high-risk and good 46 low-risk) who completed the 6-month study visit, thus this is the total number of mothers who completed the exit survey. One survey was completed per mother/infant dyad.
Measure: Count of Participants; unit: Participants
Arm/Group | High-risk Mothers | Low-risk Mothers
Number analyzed (Participants) | 7 | 46
Participants
  Testing for Mothers | 7 | 41
  Testing for Infants | 7 | 40

2. Primary Outcome: Number of Mothers With Infant Vaccination Acceptability Survey Scores >80%
Description: The acceptability of the intervention approach to participants will be defined as >80% acceptability on a single question measured using a 5-point Likert scale (range 1-5, highest score of 5 representing the highest acceptability). For example, the options for responses will include: "Very unacceptable" (1), "Somewhat unacceptable" (2), "No opinion" (3), "Somewhat acceptable" (4), "Very acceptable" (5) and "Did not allow study personnel to vaccinate my infant". Scores equal to or greater than 4 considered 80%.
Time Frame: Upon completion of the exit survey, or up to 12 months
Population: There were a total of 53 mothers (7 high-risk and 46 low-risk) who completed the 6-month study visit, thus this is the total number of mothers who completed the exit survey. One survey was completed per mother/infant dyad.
Measure: Count of Participants; unit: Participants
Arm/Group | High-risk Mothers | Low-risk Mothers
Number analyzed (Participants) | 7 | 46
Participants | 7 | 42

3. Secondary Outcome: Number of Infants With HBV Positivity at 6 Months of Life to Indicate Mother-to-Child Transmission of HBV
Description: Mother-to-child transmission of HBV is defined as HBsAg positivity in the infant at 6 months of life.
Time Frame: Measured at 6 months after birth
Population: A total of 88 infants were born to mothers in the study, but only 53 infants (7 born to high-risk mothers and 46 born to low-risk mothers) were followed through 6 months of life and tested for HBsAg at that time.
Measure: Count of Participants; unit: Participants
Arm/Group | Infants Born to High-risk Mothers | Infants Born to Low-risk Mothers
Number analyzed (Participants) | 7 | 46
Participants | 0 | 0

4. Secondary Outcome: Number of Mothers With High-risk HBV Demonstrating Adherence to Tenofovir Therapy
Description: Adherence to tenofovir therapy is defined as <20% of pills remaining on monthly pill counts for high-risk mothers with HBV receiving tenofovir
Time Frame: Pill counts to be measured monthly. Total adherence averaged over 6-month treatment period.
Measure: Count of Participants; unit: Participants
Groups:
- High-risk Mothers: Mothers with high-risk HBV who took tenofovir during pregnancy
Arm/Group | High-risk Mothers
Number analyzed (Participants) | 9
Participants | 9

5. Secondary Outcome: Number of Infants Receiving Timely Birth Dose Vaccination
Description: Timeliness of infant HBV vaccination is defined as >90% of infants receiving birth dose vaccine within 24 hours of life
Time Frame: Within 24 hours after birth
Measure: Count of Participants; unit: Participants
Arm/Group | Infants Born to High-risk Mothers | Infants Born to Low-risk Mothers
Number analyzed (Participants) | 9 | 79
Participants | 8 | 38

ADVERSE EVENTS:
Time Frame: The participants were monitored for adverse events over the duration of treatment (an average of 6 months for High-risk Mothers taking tenofovir therapy, and an average of 3 days or the duration of hospital stay for infants after receiving hepatitis B vaccination). Since Low-risk Mothers did not receive a study intervention, adverse event data was not overtly sought unless self-reported by participant.
Arm/Group | High-risk Mothers | Low-risk Mothers | Infants Born to High-risk Mothers | Infants Born to Low-risk Mothers
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/81 | 0/9 | 1/79
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/81 | 0/9 | 0/79
Other Adverse Events (participants affected / at risk) | 2/10 | 0/81 | 0/9 | 0/79
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-risk Mothers (N=10) | Low-risk Mothers (N=81) | Infants Born to High-risk Mothers (N=9) | Infants Born to Low-risk Mothers (N=79)
Rebound elevation of ALT and HBV DNA after discontinuation of Tenofovir (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — ALT = alanine aminotransferase DNA = deoxyribonucleic acid

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT03567382/Prot_SAP_000.pdf